CLINICAL TRIAL: NCT05949385
Title: A Study to Assess the Effect of Itraconazole Capsules on the Pharmacokinetics of ZX-7101A Tablets in Healthy Adult Subjects in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Zenshine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZX-7101A-205
Record Dates: First submitted 2023-06-13; First posted 2023-07-18 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Pharmacokinetics
Keywords: DDI
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ZX-7101A and Itraconazole (Experimental): D1 and D31 Take ZX-7101A tablet 40mg (1 tablet, 40mg/ tablet）,oral，fasting； D26-D50 Itraconazole capsule 200mg(2 capsules, 100mg/ capsule) ，oral in 30min after breakfast.
  Interventions: Drug: ZX-7101A

INTERVENTIONS:
Drug: ZX-7101A — Single dose of oral administration of ZX-7101A and Multiple dose of oral of Itraconazole Capsules
  Other Names: Itraconazole

SUMMARY:
The primary objective of the study is to evaluate the effect of Itraconazole on pharmacokinetics of ZX-7101 in healthy Chinese adult subjects after oral administration of ZX-7101A tablets.

The secondary objective of the study is to evaluate the safety and tolerability of single dose of ZX-7101A orally in healthy subjects.

Evaluate the effect of Itraconazole on pharmacokinetics of pre-drug ZX-7101A in healthy Chinese adult subjects after oral administration of ZX-7101A tablets.

DETAILED DESCRIPTION:
ZX-7101A tablets 40 mg once on Day 1 and Day 31, Itraconazole 200 mg once daily (QD) from Study Day 26 - 50

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between the ages of 18 and 45 years (including the threshold value, based on the date of signing ICF).
* Weight: Male weight ≥50 kg, female weight ≥45 kg, BMI between 19.0 and 28.0 kg/m2 (including cut-off value), BMI= weight (kg)/height 2 (m2).
* The investigator judged the subjects to be in good overall health based on their medical history, physical examination, vital signs, 12-lead electrocardiogram, laboratory tests (routine blood work, urine work, blood biochemistry, coagulation function), viral serology, and chest X-ray results (normal or abnormal test results have no clinical significance).
* Fertile female subjects or male subjects who voluntarily signed ICF should be no fertile, sperm/egg donation for 6 months (female) or 90 days (male) from the beginning to the last dose, and voluntary use highly effective contraception (including partner) (non-drug contraception is required during the trial).
* Fully understand the trial content and possible adverse reactions, have the ability to communicate with researchers normally, while complying with study requirements, follow protocol procedures and restrictions, and be able to visit on time.

Exclusion Criteria:

* Subjects with a prior or present history of clinically abnormal metabolic, liver, kidney, hematological, pulmonary, cardiovascular, gastrointestinal, urinary, endocrine, neurological, or psychiatric disease who were judged by the investigator to be unsuitable for participation in this study.
* Subjects with digestive tract disease or any condition that may affect drug absorption, such as a history of liver and gallbladder disease, gastrointestinal disease, gastrointestinal surgery (except appendectomy) or a history of chronic pancreatitis, idiopathic acute pancreatitis, or habitual diarrhea.
* Allergic constitutions (such as allergies to two or more drugs, foods, and pollen), or determined by the investigator, may be allergic to the investigational product or any component of the investigational product.
* Acute respiratory infections within 2 weeks before screening; Or have a history of fungal infection.
* For patients with abnormal vital signs (blood pressure, pulse rate, ear temperature) and clinically significant results, the abnormal values of each vital sign are:Body temperature (ear temperature) >37.5 ℃; Systolic blood pressure (recumbent) <90 mmHg or ≥140 mmHg; Diastolic blood pressure (lying) <50 mmHg or ≥90 mmHg; Pulse rate (lying position) <50 beats/min or >100 beats/min.
* QTcF interval > 450ms or < 300 ms (Fridericia's correction), or QRS>120ms. Abnormal liver function: alanyl aminotransferase (ALT) or aspartate aminotransferase (AST) higher than the upper limit of normal or serum total bilirubin (TBIL) greater than 1.5 times the upper limit of normal, who judged clinical significance by investigators.
* Subjects estimate glomerular filtration rate <90 mL/min/1.73 m2.
* Subjects virus serological test (hepatitis B virus surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, treponema pallidum specific antibody TPPA) positive results.
* Subjects with a history of drug abuse (morphine, dimethylene dioxyamphetamine, methamphetamine, THC, ketamine, cocaine) or who screened positive for drug abuse.
* Women who are pregnant or breastfeeding, or who test positive for blood pregnancy.
* Subjects who have used any P-gp or CYP inducer or inhibitor within 30 days before screening, or any prescription or Chinese herbal medicine within 4 weeks before the start of the trial, or over-the-counter or health care products (including polyvalent cations and metal supplements, etc.) within 2 weeks before the start of the trial; It should have a longer time interval if the elimination half-life is longer-at least 5 elimination half-lives for the drug.
* Subjects who consumed more than 14 units of alcohol per week in the 6 months prior before screening (1 unit of alcohol =360mL beer or 45mL spirits with 40% alcohol or 150mL wine) or had a positive alcohol breath test or could not abstain during the trial.
* Subjects who smoked more than 5 cigarettes per day in the 3 months prior before screening or habitually used nicotine-containing products or could not give up during the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-07-02 (Actual); Primary Completion 2023-09-23 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
PK parameters of active metabolite ZX-7101after a single oral ZX-7101A tablet and combined with multiple oral itraconazole capsules in healthy Chinese adult subjects | Day1-Day20, Day31-Day50
  Cmax
PK parameters of active metabolite ZX-7101after a single oral ZX-7101A tablet and combined with multiple oral itraconazole capsules in healthy Chinese adult subjects | Day1-Day20, Day31-Day50
  AUC0-t
PK parameters of active metabolite ZX-7101after a single oral ZX-7101A tablet and combined with multiple oral itraconazole capsules in healthy Chinese adult subjects | Day1-Day20, Day31-Day50
  AUC0-inf

SECONDARY OUTCOMES:
Rate of AE | Day1-Day20, Day31-Day50
  Rate of TEAE
PK parameters of prodrug ZX-7101A | Day1-Day20, Day31-Day50
  Cmax
PK parameters of prodrug ZX-7101A | Day1-Day20, Day31-Day50
  AUC0-t
PK parameters of prodrug ZX-7101A | Day1-Day20, Day31-Day50
  AUC0-inf
PK parameters of ZX-7101 | Day1-Day20, Day31-Day50
  Tmax
PK parameters of ZX-7101 | Day1-Day20, Day31-Day50
  CL/F

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No